CLINICAL TRIAL: NCT07292298
Title: Phase 2 Single-Arm Rectal Cancer Brachytherapy for Patients With Low-Lying Residual Adenocarcinoma After Total Neoadjuvant Therapy to Improve Organ Preservation Rates
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-1202.cc
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Rectal Adenocarcinoma; Rectal Cancer
Keywords: Locally Advanced Rectal Cancer; Non-metastatic Rectal Cancer; Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HDR Rectal Brachytherapy Boost (Experimental): The intervention consists of a boost using Iridium-192 delivered via an intracavitary applicator in three weekly fractions totaling 21 Gy. The goal is to improve organ preservation rates and avoid surgical resection (APR or low LAR). Treatment planning includes MRI, endoscopic clip placement, and CT simulation prior to each fraction.
  Interventions: Radiation: High Rare Dose Rectal Brachytherapy Boost

INTERVENTIONS:
Radiation: High Rare Dose Rectal Brachytherapy Boost — HDR rectal brachytherapy boost using Iridium-192 delivered via an intracavitary applicator in three weekly fractions (total dose: 21 Gy) for patients with low-lying residual rectal adenocarcinoma following total neoadjuvant therapy.

SUMMARY:
Rectal cancer patients who do not achieve a complete response to standard of care chemotherapy and radiation often require surgical resection as part of curative intent therapy. This study will evaluate whether additional "focal" radiation delivered internally (rectal brachytherapy) can provide complete responses and thus spare the requirement for surgery.

The main questions are whether: 1) rectal brachytherapy is safe in this clinical treatment paradigm and if 2) rectal brachytherapy improves organ preservation (no need for surgery).

The trial involves an additional MRI pelvis and sigmoidoscopy with marker placement to define high-risk residual disease for radiation planning. Subsequently, 3 outpatient brachytherapy treatments are given on a weekly basis. If a patient achieves a complete response to brachytherapy, standard of care non-operative surveillance visits are conducted with study visits aligned during the first two years following brachytherapy.

DETAILED DESCRIPTION:
Rectal cancer patients with incomplete responses following standard of care chemotherapy and radiation are offered surgery as part of curative intent regimens. Similarly, patients with near-complete responses following initial therapy may require future salvage surgery given high local recurrence risk in the rectum. The goal of this study is to determine whether additional "internal" focal radiation delivered by rectal brachytherapy can provide a complete tumor response, such that patients can avoid surgical intervention. While rectal brachytherapy efficacy, technique, and safety has been demonstrated in previous studies conducted in Europe and Canada, it has not been tested to "boost" responses following standard of care chemotherapy/radiation in the United States.

Specifically, rectal brachytherapy treatment requires placement of a multichannel cylinder into the rectum following local analgesia and oral medication to improve procedure tolerability. A balloon on the cylinder is inflated to displace rectum uninvolved with tumor away from the internal high-dose radiation source that travels through the cylinder channels abutting the tumor. 21 Gy cumulative dose over 3 weekly treatments is administered to the high-risk rectal mucosa at a depth aligning to tumor thickness. The cylinder will be immobilized in the rectum for up to 3 hours during each of the 3 brachytherapy sessions, with radiation treatment being less than 10 minutes following completion of planning.

If complete response is achieved, surveillance visits will be conducted with an almost identical protocol to patients who achieve complete response following standard of care radiation/chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Adults (18-100 years old)
4. ECOG 0-3
5. Patients with MMR-proficient low-mid rectal adenocarcinoma cT1-4 N0-2 M0 who underwent total neoadjuvant therapy who have not achieved complete response (i.e. incomplete or near-complete) in the rectal primary tumor such that surgical resection, if offered presently or in the future, would be an APR or low LAR per colorectal surgeon expert opinion and central review at University of Colorado rectal tumor board. Tumor restaging will be 4-16 weeks following completion of total neoadjuvant therapy, and no sooner than 8 weeks if patients received chemotherapy followed by chemoradiation/short course radiation.
6. Residual rectal disease must have its craniocaudal extent <4 cm with thickness <1.2 cm. Tumor must have <50% circumferential involvement. Residual disease must be above the dentate line and not involving the anal canal.
7. In patients with original cN1-2 disease, restaging CT and MRI after total neoadjuvant therapy must demonstrate at least near-complete response of the pelvic lymph nodes per NCCN criteria as evaluated by central review at University of Colorado rectal tumor board.
8. Interval of time between completion of TNT and initiation of rectal brachytherapy must be between 4-16 weeks.
9. Patients must be recovered from total neoadjuvant therapy and must not have significant rectal incontinence at time of screening.
10. Received conventionally fractionated external beam chemoradiation between 45-56 Gy or short-course external beam radiation prescription of 25 Gy to rectal mucosa, in addition to systemic chemotherapy before or after radiation per National Comprehensive Cancer Network (NCCN) guidelines.
11. Women of child-bearing potential must have a negative urine or serum pregnancy test within 14 days of HDR treatment.
12. Men and women of reproductive potential who are sexually active must agree to follow instructions of contraception for the duration of the study and 6 months post-rectal brachytherapy completion.
13. CBC at the time of screening must have platelets>50 10^9/L, Hemoglobin>8 g/dL and Absolute Neutrophil Count > 500 10^9/L

Exclusion Criteria:

1. History of ulcerative colitis or Crohn's disease.
2. Pelvic radiotherapy given prior to rectal cancer external beam radiation.
3. Prior colorectal surgery in which anastomotic site is at or near HDR brachytherapy target.

   o Prior local excision is not an exclusion criterion.
4. Uncontrolled intercurrent severe illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
5. Life expectancy <3 years per provider discretion.
6. Concurrent administration of any cytotoxic chemotherapy, immunotherapy, or other any targeted oncologic agent that would impact rectal cancer is not allowed during study protocol.
7. If rectal cancer has been treated outside of standard total neoadjuvant therapy per NCCN guidelines, patients are ineligible for the trial. This includes if patients received external beam chemoradiation dose with prescription >56 Gy or short-course radiation to rectal mucosa prescription >30 Gy.
8. Pregnant women.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-11 (Estimated); Primary Completion 2030-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Organ preservation (no surgical requirement) of the rectum associated with complete clinical response | 2 years following study treatment
  As evaluated by standard of care sigmoidoscopy and MRI

SECONDARY OUTCOMES:
Locoregional recurrence free survival | 2 years following study treatment
  As defined by CT and MRI pelvis
Distant metastatic free survivial | 2 years following study treatment
  As assessed by CT c/a/p
Overall survival | 2 years following study treatment
  Overall survival
Bowel function | 2 years following study treatment
  As assessed by LARS (low anterior resection syndrome) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David Binder, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Rochester Medical Center, Rochester, New York
  - Oregon Health and Sciences University, Portland, Oregon